CLINICAL TRIAL: NCT00716001
Title: Effect of Hydration With Sodium Bicarbonate for Long-Term Clinical Outcomes in Patients With Chronic Kidney Disease Undergoing an Emergent Coronary Procedure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Osaka General Medical Center (Other)
Responsible Party: Masaharu Masuda, Osaka General Medical Center
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: OPTSB
Record Dates: First submitted 2008-07-02; First posted 2008-07-15 (Estimated); Last update posted 2008-07-15 (Estimated); Status verified 2008-07

CONDITIONS: Chronic Renal Failure
Keywords: patients with chronic renal failure undergoing elective percutaneous coronary intervention
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NAC (Active Comparator)
  Interventions: Drug: N-acetylcysteine
- nonNAC (Placebo Comparator)
  Interventions: Drug: N-acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine

SUMMARY:
This study is to evaluate the efficacy of sodium bicarbonate plus N-acetylcysteine for the prevention of contrast-induced nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic renal failure(serum creatinine >1.1mg/dl) undergoing elective percutaneous coronary intervention

Exclusion Criteria:

* administered with sodium bicarbonate and/or N-acetylcysteine and/or contrast media within 72 hours.
* pregnancy
* congestive heart failure
* allergy to sodium bicarbonate and/or N-acetylcysteine
* hemodialysis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2008-07; Primary Completion 2009-06 (Estimated)